CLINICAL TRIAL: NCT06682247
Title: A Real-world Study of Chidamide in Combination with PD-1/PD-L1 Antibodies and Anti-angiogenic Agents in the Treatment of Microsatellite Stable Advanced Colorectal Cancer
Brief Title: A Real-world Study of Chidamide in Combination with PD-1/PD-L1 Antibodies and Anti-angiogenic Agents in Advanced MSS Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Feng Wang (Other)
Responsible Party: Sponsor-Investigator, Feng Wang, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: CSIIT-Q88
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Bevacizumab; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- chidamide + PD-1/PD-L1 inhibitors +Bevacizumab or tyrosine kinase inhibitors
  Interventions: Drug: Chidamide, Tucidinostat; PD-1/PD-L1 inhibitor or double antibodies; Bevacizumab or tyrosine kinase inhibitors

INTERVENTIONS:
Drug: Chidamide, Tucidinostat; PD-1/PD-L1 inhibitor or double antibodies; Bevacizumab or tyrosine kinase inhibitors — Chidamide, Tucidinostat; PD-1/PD-L1 inhibitor or double antibodies; Bevacizumab or tyrosine kinase inhibitors

SUMMARY:
This is an observational , multicenter, real-world study aimed at evaluating the efficacy and safety of the combination of immune checkpoint inhibitors, chidamide and antiangiogenic agents in Microsatellite Stable advanced colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years
2. Histology-confirmed metastatic CRC (mCRC);
3. ECOG 0~2
4. At least one efficacy evaluation
5. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Lack of follow-up data.
2. Chidamide stopped after less than two cycles.
3. Serious comorbidities that interfere with the efficacy or safety analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced/metastatic MSS colorectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 years

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
Clinical Benefit Rate (CBR) | 2 years
Disease Control Rate （DCR） | 2 years
Overall survival (OS) | 2 years